CLINICAL TRIAL: NCT03844282
Title: Research Evaluating Sports ConcUssion Events - Rapid Assessment of Concussion and Evidence for Return
Acronym: RESCUE-RACER
Status: Completed | Type: Observational
Sponsor: University of Cambridge (Other)
Collaborators: Global Institute for Motorsport Safety (GIMSS) - Year 1 (Unknown); Neurolign Technologies LLC (previously Neuro Kinetics Incorporated, NKI) (Unknown); Cambridge University Hospitals NHS (National Health Service) Foundation Trust (Unknown); Federation Internationale de l'Automobile - Year 2 onwards (Unknown)
Responsible Party: Principal Investigator, Naomi D Deakin, Study Coordinator, University of Cambridge
Other Study IDs: A094577
Record Dates: First submitted 2018-11-12; First posted 2019-02-18 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Concussion, Brain; Motor Vehicle Accident
Keywords: Concussion; mTBI; mild traumatic brain injury; motorsport; motor sport; racing
MeSH Terms: conditions — Brain Concussion | interventions — Neuropsychological Tests; Vision, Ocular; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Saliva will be collected from RESCUE-RACER participants during each study visit or assessment. All saliva samples will be centrifuged to render them acellular, therefore ensuring that they are no longer relevant material as defined by guidance from the United Kingdom (UK) Human Tissue Authority (see https://www.hta.gov.uk/policies/list-materialsconsidered-be-%E2% 80%98relevant-material%E2%80%99-under-human-tissue-act-2004).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- CArBON (baseline): The RESCUE-RACER programme is formed of two studies; baseline (CArBON) and one post-injury (CARS). At baseline the larger CArBON study involves completion of a thorough single baseline neuroscientific assessment of healthy motorsport competitors including clinical, neuropsychological, neurocognitive, biomarker and vestibulo-ocular assessments, in addition to MRI of the brain.
  Interventions: Diagnostic Test: Clinical assessment (SCAT5); Diagnostic Test: ImPACT; Behavioral: CANTAB; Diagnostic Test: I-PAS/Dx100; Biological: Saliva sample; Other: fMRI
- CARS (exposure to a potentially concussive event): The RESCUE-RACER programme has a single post-injury study; after involvement in a potentially concussive event sustained during motorsport, CARS serially repeats the CArBON assessment battery in the immediate post-concussion recovery period. CARS participants will under-go post-exposure neuroscientific assessments immediately after injury and then at one, two and three weeks post-injury. If symptoms persist beyond this time, a further two assessments at monthly intervals will be offered.
  Interventions: Diagnostic Test: Clinical assessment (SCAT5); Diagnostic Test: ImPACT; Behavioral: CANTAB; Diagnostic Test: I-PAS/Dx100; Biological: Saliva sample; Other: fMRI

INTERVENTIONS:
Diagnostic Test: Clinical assessment (SCAT5) — The SCAT5 is a standardized tool for evaluating sports-related concussions designed for use by physicians and licensed healthcare professionals in patients aged 13 years and above. It is a ten minute paper-based assessment which includes immediate and office/off-field assessments. SCAT5 incorporates the Maddocks' questions, Glasgow Coma Scale (GCS), cervical spine assessment and symptom evaluation, in addition to cognitive and neurological screening.
  Other Names: Sports Concussion Assessment Tool 5
Diagnostic Test: ImPACT — ImPACT (Immediate Post-Concussion Assessment and Cognitive Testing) is a neurocognitive assessment administered online or using desktop software in a controlled environment. ImPACT has two components: baseline testing and post-injury testing, both of which are used to determine if a patient can safely return to sporting activity post-concussion.
  Other Names: Immediate Post-concussion Assessment and Cognitive Testing; ImPACT concussion test
Behavioral: CANTAB — Originally developed at the University of Cambridge, the Cambridge Neuropsychological Test Automated Battery (CANTAB) platform includes highly sensitive, precise and objective measures of cognitive function, correlated to neural networks. These tests have demonstrated sensitivity to detecting changes in neuropsychological performance and include tests of working memory, learning and executive function; visual, verbal and episodic memory; attention, information processing and reaction time; social and emotion recognition, decision making and response control.
  The CANTAB touchscreen battery (www.camcog.com) will be utilised to perform neuropsychological assessments within RESCUE-RACER, whose study-specific protocol may include assessments of: Spatial Working Memory (working memory and strategy), Reaction Time (processing and psychomotor speed), Paired Associated Learning and the Multi-Tasking Test.
  Other Names: CANTAB Connect; Cambridge Cognition CANTAB battery; CANTAB battery
Diagnostic Test: I-PAS/Dx100 — I-PAS™ (now re-named Dx 100) is a portable, head-mounted, neural functional assessment tool. With its integrated clinical eye tracking and digital display, the FDA has cleared (K171884) fourteen tests and an unmatched list of variables for clinical use for a variety of conditions. This utility of this device will be investigated for motorsport-related concussion.
  Other Names: OVRT; Ocular, vestibular and reaction time testing; I-Portal Portable Assessment System; Video Oculography; Dx100
Biological: Saliva sample — Micro RNA's (miRNA's) are easily measured in saliva and have proven to have both diagnostic and prognostic use in sports-related concussion across the adolescent and adult populations, with levels persisting for some weeks after the concussive event. RESCUE-RACER will collect saliva samples for analysis of biomarkers of concussion, which may include miRNA and other markers of injury.
Other: fMRI — RESCUE-RACER participants will be invited to complete a functional MRI scan, whose 90-minute protocol may include: multi-parametric mapping (MPM), susceptibility weighted imaging (SWI), diffusion weighted imaging (DWI), proton spectroscopy and functional MRI (fMRI) with blood oxygenation-level dependent contrast (BOLD), completed at 7T (Tesla), or 3T if this is not possible.
  Other Names: Magnetic Resonance Imaging; Function MRI

SUMMARY:
RESCUE-RACER is jointly sponsored by the University of Cambridge and Cambridge University Hospitals NHS Foundation Trust.

The RESCUE-RACER programme evaluates motorsports competitors at baseline (CArBON) and post-injury (CARS). The CArBON study (Competitor Assessment at Baseline; Ocular, Neuroscientific) collects a battery of neuroscientific data in a baseline assessment. The CARS study (Concussion Assessment and Return to motorSport), repeats the CArBON battery throughout the recovery period in competitors who sustain a potentially concussive event during motorsport.

The primary outcome of the RESCUE-RACER programme is to establish the natural history of concussive symptoms and signs in motorsport competitors using a comprehensive neuroscientific battery. The standard clinical assessment of concussive symptoms will be correlated with objective clinical scoring, in addition to neurocognitive and neuropsychological assessments. Advanced brain imaging with MRI will be used to further characterize head injuries in motorsport. Finally, salivary biomarkers will be collected to monitor the measurable biological effects of a potentially concussive event immediately following injury and through recuperation in the recovery period.

The secondary outcome is investigation of a novel diagnostic tool for concussion, in the form of a 3D head-mounted display and eye tracking system capable of assessing ocular, vestibular and reaction time (OVRT) functions (the I-PAS device, now re-named Dx 100).

The results of RESCUE-RACER will form an evidence base for medical decision-making track side after a potentially-concussive incident and will advise on clinic management of motorsports concussion, including the important 'return-to-race' decision.

ELIGIBILITY:
Inclusion criteria (CArBON and CARS)

a) Competitive motorsports participants

Additional inclusion criteria - CARS only

1. Exposure to a potentially concussive event during motorsport activity OR a diagnosis of concussion during motorsport made by an experienced clinician <3 weeks prior to referral.
2. Mental capacity to consent to study participation

Exclusion criteria (CArBON) Prior severe or moderate traumatic brain injury, diagnosis of mild traumatic brain injury or concussion within the last 6 months, symptoms of head injury at time of enrolment

Exclusion criteria - (CArBON and CARS)

Absolute exclusion criteria

1. Age <16 years
2. Ongoing injuries so severe as to preclude study enrolment
3. Recent (within the last 4 months) or current involvement in a research study involving administration of trial medication

Possible exclusion criteria i. Recent (within the last 4 months) or current involvement in an observational research study (decision made by the enrolling study team member based upon the study's time commitments and the likelihood and feasibility of the participant attending future RESCUE-RACER assessments) ii. For MRI imaging only; metal implants or exposure to metal foreign objects (such as welding) - as per local policy (at the University of Cambridge Wolfson Brain Imaging Centre, WBIC).

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Eligibility Criteria-CArBON; all competitors associated with the TOCA* series or contracted by Aston Martin Racing (AMR)
  Eligibility Criteria-CARS; following exposure to a potentially concussive event sustained during motorsport activity: a) All competitors associated with the TOCA series or contracted by AMR b) Any competitive motorsports competitors who are referred to the Chief Investigator
  *'TOCA' is a motorsports event package based in the UK (registered as a Patient Identification Centre, PIC). In 2019, TOCA consists of 6 semi-/professional racing series (3 adult-British Touring Car Championship (BTCC), Porsche Carrera Cup GB, Michelin Ginetta GT4 Supercup; 1 mixed age-Renault UK Clio Cup (17 years+); 2 adolescent (14-17 years)-Simpson Race Products Ginetta Junior Championships, British Formula 4 Championship; certified by Fédération Internationale de l'Automobile, FIA; powered by Ford).In 2020, Renault is replaced by the Mini Challenge series.
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2018-11-09 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change in SCAT5 decision scores | Baseline (CArBON assessments) to 1-3 weeks after concussion (CARS assessments)
  Change in performance on the Sports Concussion Assessment Tool 5 (SCAT5) from baseline to follow-up, as measured by sections of the assessment:
  1. Symptoms - number (range 0-22) and severity (each rated as 0-6), summed to form a symptom severity score (range 0-132), with higher scores indicating worse symptoms *For more information please see Step 2: Symptom Evaluation at link below*
  2. Orientation score
  3. Immediate memory score
  4. Concentration score
  5. Neurological examination
  6. Number of balance errors
  7. Delayed recall score
  Which are combined to form a Decision (please see Step 6 at https://bjsm.bmj.com/content/bjsports/early/2017/04/26/bjsports-2017-097506SCAT5.full.pdf).
Change in computerised neurocognitive assessment scores | Baseline (CArBON assessment) to 1-3 weeks after concussion (CARS assessments)
  Change in neurocognitive performance from baseline to follow-up, as measured by the Immediate Post-concussion Assessment and Cognitive Testing tool (ImPACT, please see https://impacttest.com/).
  This previously-validated assessment consists of the following sections:
  1. Attention (including processing)
  2. Memory (verbal and visual recognition; visual working)
  3. Visual motor speed
  4. Learning
  5. Impulse control (response inhibition)
  6. Delayed memory (repeat of verbal and visual tasks in 2)
  Which are combined to form Composite scores, whose calculation is defined in the ImPACT's Administration & Interpretation Manual (available on request).
Change in computerised neuropsychological assessment scores | Baseline (CArBON assessment) to 1-3 weeks after concussion (CARS assessments)
  Change in neuropsychological performance from baseline to follow-up, as measured by CANTAB Connect Research, the world's most validated, precise and reliable research software (please see http://www.cambridgecognition.com/products/cognitive-research/).
  This previously-validated assessment software consists of the following sections:
  1. Attention (processing and psychomotor speed)
  2. Memory (visual episodic)
  3. Executive function and decision-making (working memory and strategy; planning).
  Each assessment produces a number of outputs, as detailed in the CANTAB Connect Research Overview Document (available on request).
Change in the brain's microstructural architecture, or functional changes in the brain | Baseline (CArBON assessment) to 1-3 weeks after concussion (CARS assessments)
  Change in the brain's microstructural architecture, or functional changes in the brain, from baseline to follow-up as measured by:
  1. High-resolution structural imaging - disruption of usual cerebral architecture (i.e. volume of sub/cortical structures)
  2. Susceptibility-weighted imaging (SWI) - signal alteration
  3. Diffusion-weighted imaging (DWI) - voxel intensity
  4. Resting-state functional MRI (fMRI) - changes in blood oxygenation level
  5. Proton spectroscopy
Change in salivary biomarker levels | Baseline (CArBON assessments) to 1-3 weeks after concussion (CARS assessments)
  Change in the levels of salivary biomarkers from baseline to follow-up as potentially measured by markers of:
  1. Neuronal injury - such as neurofilament light chain (NFL)
  2. Glial injury - such as S100B (a calcium-binding peptide)
  3. Epigenetic effects - as measured by micro RNA levels (miRNA)
  4. Neurofibrillary degeneration - as measured by tau.

SECONDARY OUTCOMES:
Altered performance in ocular, vestibular and reaction time (OVRT) assessment utilising the I-PAS/Dx100 device | Baseline (CArBON assessments) to 1-3 weeks after concussion (CARS assessments)
  The applicability of OVRT assessment as a diagnostic tool for motorsport concussion will be investigated by correlating changes in OVRT performance at baseline to OVRT performance following a clinical diagnosis of concussion or participation in motorsport activity. The assessment will be conducted with a portable head-mounted 3D display (please see http://neurolign.com/our-technology/, previously https://www.neuro-kinetics.com/products/).
  Alteration in OVRT performance will be measured using:
  1. Ocular tests - saccades (vertical, horizontal, predictive, self-paced, memory-guided and anti-), smooth pursuit, optokinetic reflex, vergence, light reflex
  2. Vestibular tests - subjective visual vertical
  3. Reaction time assessments - auditory, visual
  The I-PAS/Dx100 training manual is available on request (publication of further assessment details is subject to patents and/or copyright).

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Hutchinson, MB BS FRCS (Surg Neurol), Principal Investigator — University of Cambridge
Locations (1):
- Mr Stephen Kelleher, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
As per University of Cambridge and Cambridge University Hospitals, CUH, protocol, study data may be accessed by members of relevant clinical or research teams. A summary of anonymised aggregated data collected each year will be shared with the Funder in the form of an annual report. Linked and robustly anonymised OVRT data will be encrypted and electronically shared with collaborators at Neuro Kinetics Incorporated (now Neurolign) for the purpose of analysis, subject to a Data Transfer agreement approved by Cambridge University Hospitals (CUH, joint co-sponsor). Transfer of this study data will be in accordance with Health Research Authority (HRA) guidance 'Sharing of Anonymous Data Collected for Research Purposes'.
Supporting Information: Study Protocol, ICF
Time Frame: CArBON data will be available following agreement of the report by all collaborators (estimated to be late 2020); CARS data will be handled in the same way (estimated middle of 2021).
Access Criteria: Data will only be made available to collaborators, subject to the programme's research agreement.

REFERENCES:
- [Derived] Deakin ND, Suckling J, Hutchinson PJ. Research Evaluating Sports ConcUssion Events-Rapid Assessment of Concussion and Evidence for Return (RESCUE-RACER): a two-year longitudinal observational study of concussion in motorsport. BMJ Open Sport Exerc Med. 2021 Jan 13;7(1):e000879. doi: 10.1136/bmjsem-2020-000879. eCollection 2021. PMID 33500784
- See also: RESCUE-RACER study website — http://www.rescueracer.org
- See also: RESCUE-RACER Twitter account — https://twitter.com/rescue_racer
- See also: RESCUE-RACER Facebook account — https://www.facebook.com/RESCUERACER
- See also: RESCUE-RACER Instagram account — https://www.instagram.com/rescue_racer/
- See also: RESCUE-RACER published study protocol — https://bmjopensem.bmj.com/content/7/1/e000879

DOCUMENTS (1):
  • Informed Consent Form (2018-08-28): https://cdn.clinicaltrials.gov/large-docs/82/NCT03844282/ICF_002.pdf